CLINICAL TRIAL: NCT06392074
Title: A Randomized, Double-blind, Three-part, Two-period, Two-sequence, Single-dose, Cross-over Study to Compare the Pharmacokinetics (PK), Safety and Immunogenicity Profile of MB04 (Proposed Etanercept Biosimilar), EU-sourced Enbrel® and US Licensed Enbrel® in Healthy Male Volunteers
Brief Title: A Study Investigating the Safety, Absorption, and Elimination of MB04, a New Compound That May Potentially be Used in the Treatment of Autoimmune Disorders
Acronym: MB04-A-01-23
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB04-A-01-23
Record Dates: First submitted 2024-03-11; First posted 2024-04-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — etanercept biosimilar SB4; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MB04 (etanercept biosimilar) (Experimental): 1 mL pre-filled single-use syringe containing 50 mg (50mg/mL) of etanercept
  Interventions: Drug: MB04
- US licensed Enbrel (etanercept) (Active Comparator): 1 mL pre-filled single-use syringe containing 50 mg (50mg/mL) of etanercept
  Interventions: Drug: US License Enbrel
- EU sourced Enbrel (etanercept) (Active Comparator): 1 mL pre-filled single-use syringe containing 50 mg (50mg/mL) of etanercept

INTERVENTIONS:
Drug: MB04 — Subcutaneous injection
  Other Names: (etanercept biosimilar)
  Arms: MB04 (etanercept biosimilar)
Drug: US License Enbrel — Subcutaneous injection
  Other Names: (etanercept)
  Arms: US licensed Enbrel (etanercept)
Drug: EU Source Enbrel — Subcutaneous injection
  Other Names: (etanercept)

SUMMARY:
This is a randomized, double-blind, three-part, two-sequence per part, two-period, single-dose, cross-over study in healthy male volunteers to compare the PK, safety, and immunogenicity of MB04 and EU /US Enbrel®.

During the course of the study, the similarity in pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms. Safety, tolerability, and immunologic response to the administered drugs will also be evaluated throughout.

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate PK similarity between MB04 and EU-Enbrel®, between MB04 and US Enbrel® as well as between EU-Enbrel® and US-Enbrel®. Additional PK parameters will be evaluated as secondary endpoints.

Safety and tolerability will be assessed through Adverse Events, clinical laboratory, vital signs, ECGs, and physical examination findings, and any other parameter that is relevant for safety assessment.

The incidence of ADA to etanercept and the neutralizing potential and titre of positive ADA will be reported

ELIGIBILITY:
Inclusion Criteria

1. BMI: 18.5 kg/m2 to 29.9 kg/m2, inclusive, at screening.
2. Weight: ≥60 kg to ≤100 kg, inclusive, at screening.
3. Status: healthy subjects.
4. Male subjects, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from first admission to the clinical research center until 3 months after the last study drug administration. Adequate contraception for the male subject (and his female partner, if she is of childbearing potential) is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm, a cervical cap, or a condom. Total abstinence from heterosexual intercourse, in accordance with the lifestyle of the subject, is also acceptable.
5. Ability and willingness to abstain from alcohol from 48 hours (2 days) prior to each study visit to the clinical research center.
6. Ability and willingness to abstain from methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks) and grapefruit (juice) from 48 hours (2 days) prior to each study visit to the clinical research center.
7. No presence of any clinically relevant abnormality identified by a detailed medical history and no clinically significant abnormal findings during screening, clinical examination, laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is acceptable), vital signs, and 12-lead ECG.
8. Able to comprehend and willing to sign an ICF and to abide by the study restrictions. Subjects must have signed the ICF before any study-related procedure or evaluation is performed.

Exclusion Criteria

1. Previous participation in the current study.
2. Employee of ICON or the Sponsor.
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
4. Previous exposure to the study drug (etanercept).
5. History of sensitivity to latex.
6. History or presence of any disease or condition clinically relevant which might compromise the hemopoietic, renal, hepatic, endocrine, pulmonary (in light smokers, no signs or symptoms of chronic bronchitis: sputum, recurrent bronchitis or bronchospasm), central nervous, autonomic nervous, cardiovascular, immunological, dermatological, gastrointestinal, or any other body system or psychiatric disorder, as determined by the Investigator.
7. Any current or recent history of active infections, including localized infections (within 2 months prior to the screening visit for any serious infection which requires hospitalization or intravenous (IV) anti infective, and within 14 days prior to the screening visit for known coronavirus disease 2019 (COVID-19) infection (positive antigen or polymerase chain reaction [PCR] severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] test) or any active infection which requires anti-infective oral treatment).
8. History of tuberculosis (latent or active); have a positive QuantiFERON-TB Gold test during screening (if QuantiFERON-TB Gold test result is indeterminate, the subject will not be enrolled in this study).
9. Have the intention to travel to regions where tuberculosis and mycosis are endemic diseases within 3 months after dosing.
10. Receipt of live-attenuated or live vaccine within the last 2 months before randomization or planned vaccination (live vaccines) during the study period.
11. Receipt of COVID-19 vaccine within 2 months before randomization; or plans to receive a COVID-19 vaccine within 9 weeks after study first dosing; or presence of COVID-19 symptoms within 3 weeks prior to randomization.
12. Any clinically significant laboratory finding at the time of screening.
13. A negative result for human immunodeficiency virus (HIV) and hepatitis B and C is required for participation (if the subject shows a positive hepatitis B test compatible with prior immunization and not infection, the subject may be included at the discretion of the Investigator).
14. Current malignancy or malignancy within the last 5 years (with the exception of excised non melanoma skin cancer).
15. Active smokers, or who have smoked more than 5 cigarettes a day within the last 12 months prior to start of the study and who have no signs or symptoms of chronic bronchitis.
16. All prescribed medication must have been stopped at least 30 days prior to first admission to the clinical research center.
17. All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (eg, St. John's wort) must have been stopped at least 14 days prior to first admission to the clinical research center. An exception is made for paracetamol and nonsteroidal anti-inflammatory drugs (NSAIDs), which is allowed up to admission to the clinical research center.
18. Clinically relevant history of alcoholism, addiction or drug/chemical abuse prior to screening, and/or positive alcohol and/or drug test screen confirmed by repeat at screening or check-in.
19. Donation or loss of more than 450 mL of blood within 60 days prior to the first drug administration. Donation or loss of more than 1.5 L of blood in the 10 months prior to the first drug administration in the current study.
20. Participation in a drug study within 30 days prior to the first drug administration in the current study. Participation in 4 or more other drug studies in the 12 months prior to the first drug administration in the current study.
21. Presence of tattoo or scars or any type of skin lesions at the proposed site of injection, that is interfering with the abdominal injection.
22. Subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration versus time curve (AUC) from time zero to infinity (AUC0-inf) | Day 1 to day 62
  Predose and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312, 408, and 600 h post dose
Maximum observed serum concentration (Cmax) | Day 1 to day 62
  Predose and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312, 408, and 600 h post dose

SECONDARY OUTCOMES:
AUC from time zero to the last quantifiable concentration (AUC0-last) | Day 1 to day 62
  Predose and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312, 408, and 600 h post dose
Time to reach Cmax (tmax) | Day 1 to day 62
  Predose and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312, 408, and 600 h post dose
Total body clearance (CL/F) | Day 1 to day 62
  Predose and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312, 408, and 600 h post dose
Terminal half-life (t½) | Day 1 to day 62
  Predose and at 6, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 312, 408, and 600 h post dose
Incidence of anti-etanercept antibodies (ADA) and neutralizing antibodies (Nab) | Day 1 to day 62
  Predose and, on Days 7, 14, and 26

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Clinical Research Unit, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided